CLINICAL TRIAL: NCT00304967
Title: A Study of Crystalline Proteins in Young Normal Lenses Using the NASA-NEI Dynamic Light Scattering (DLS) Device
Brief Title: Dynamic Light Scattering to Study Crystalline Proteins in Young Normal Lenses
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060117; 06-EI-0117
Record Dates: First submitted 2006-03-18; First posted 2006-03-20 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-03-31

CONDITIONS: Healthy
Keywords: Cataract; Normal Lenses; Lens Crystallines; Dynamic or Quasielastic Light Scattering (DLS); Eye Examinations; Healthy Volunteer; HV; Eye Examination
MeSH Terms: conditions — Cataract

SUMMARY:
This study will use a method called dynamic light scattering (DLS) to study the lens of the eye in young normal subjects. The DLS device uses a very dim laser light to study the lens of the eye. It detects proteins in the lens, identifying early changes that may make the device useful in future cataract studies. This study will use DLS to examine the characteristics of proteins in healthy young lenses that can be used for comparison with lenses in older people and people with cataracts.

Normal volunteers aged 5 to 21 years may be eligible for this study. Participants undergo the following procedures:

Medical history

Eye examination with dilation to include:

* Measurement of visual acuity
* Examination of pupils and eye movements
* Examination of the front of the eye (cornea, lens) with a slit lamp bio-microscope
* Examination of retina with an ophthalmoscope (instrument with a strong light and magnifying lens)
* Dynamic light scattering

DETAILED DESCRIPTION:
The NASA-NEI Dynamic Light Scattering (DLS) device detects early molecular lens changes before clinical means are able to detect any lens changes in animal and limited human studies. This ability will make it very useful in future clinical studies of cataract etiology as well as treatment. A recently concluded clinical cross sectional study of lenses (in vivo) using the DLS device showed good reproducibility and good correlation with clinical cataract grading. It also detected remarkable changes in the lens crystalline proteins with aging and with cataract formation. We therefore propose to study the characteristics of the crystalline proteins in pristine young normal lenses with DLS for comparison with aging and cataractous lens findings. We will examine 30 young normal subjects, perform undilated eye examinations, and obtain DLS measurements of their lenses. We will then use these DLS measurements for comparison with the previously obtained aging and cataract DLS measurements, to obtain normative data for future lens and cataract clinical studies.

ELIGIBILITY:
* INCLUSION CRITERIA

The study will enroll 30 normal control subjects, aged 5-21 years. Eligible participants must have normal clear lenses as determined by the eye examination.

EXCLUSION CRITERIA

Individuals who cannot cooperate or keep still for the DLS measurements will be excluded.

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30
Dates: Start 2006-03-15; Study Completion 2007-03-31

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Van Laethem M, Babusiaux B, Neetens A, Clauwaert J. Photon correlation spectroscopy of light scattered by eye lenses in in vivo conditions. Biophys J. 1991 Feb;59(2):433-44. doi: 10.1016/S0006-3495(91)82237-8. PMID 2009358